CLINICAL TRIAL: NCT05073133
Title: A Phase IV Open-label, Single-arm, Single-dose, Multicenter Study to Evaluate the saFEty, toLerability and effIcacy of Gene Replacement Therapy With intravenousOAV101(AVXS101) in Pediatric Patients From Latin America With Spinal Muscular Atrophy (SMA) - OFELIA
Brief Title: Safety and Efficacy of Intravenous OAV101 (AVXS-101) in Pediatric Patients With Spinal Muscular Atrophy (SMA) (OFELIA)
Acronym: OFELIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COAV101A1IC01; 2023-000864-67 (EudraCT Number)
Record Dates: First submitted 2021-09-20; First posted 2021-10-11 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Muscular Atrophy, Spinal
Keywords: Zolgensma; OAV101; AVXS 101; gene therapy; Muscle atrophy; SBMA; spinal and bulbar muscular atrophy; spinal muscular atrophy; bulbar muscular atrophy; muscle function; myopathy; muscle wasting; atrophied muscle; loss of muscle strength
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Atrophy; Bulbo-Spinal Atrophy, X-Linked; Muscular Diseases | interventions — Zolgensma

STUDY DESIGN:
Intervention Model Description: OAV101 will be administered as a single IV infusion at 1.1e14 vg/kg over approximately 60 minutes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OAV101 (Experimental): A single IV infusion at 1.1e14 vector genome (vg)/kg over approximately 60 minutes
  Interventions: Genetic: OAV101

INTERVENTIONS:
Genetic: OAV101 — A single Gene Therapy IV infusion at 1.1e14 vector genome (vg)/kg over approximately 60 minutes
  Other Names: AVXS-101, Zolgensma

SUMMARY:
This was a phase IV Open-label, single-arm, single-dose, multicenter study, to evaluate the safety, tolerability and efficacy of intravenous administration of OAV101 (AVXS-101) in patients with SMA with bi-allelic mutations in the survival motor neuron 1 (SMN1) gene ≤ 24 months and weighing ≤ 17 kg, over a 18-month period post infusion.

DETAILED DESCRIPTION:
This is an open-label, single arm, multi-center study to evaluate the safety, tolerability, and efficacy of IV OAV101 in symptomatic SMA pediatric participants. The study enrolled participants ≤ 24 months old that weigh ≤ 17 kg. Participants who met eligibility criteria at Screening and Baseline visits received a single dose of IV OAV101 t the approved dose of 1.1e14 vg/kg and were followed for 18 months. The study included a 20-day screening period in which there were 2 Screening visits, during which, eligibility was assessed (Screening 1), weight was collected for dose calculation (Screening 2), and baseline assessments were performed prior to treatment.

On Day -1, participants were admitted to the hospital for pre-treatment baseline procedures including prednisolone treatment per study protocol. On Day 1, participants received a single IV infusion of OAV101. Participants were discharged 12-48 hours after the infusion, based on Investigator judgment. Safety monitoring was performed on an ongoing basis per protocol requirement and was evaluated by the clinical safety team as well as DMC (Data monitoring committee).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent obtained prior to any assessment performed
2. Symptomatic SMA diagnosis based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and any copy of SMN2 gene.
3. Age ≤ 24 months of age at time of treatment

3. Weight ≤17 kg at the time of Screening Period 4. Naïve to treatment or have discontinued an approved drug/therapy 5. Up-to date on recommended childhood vaccinations and RSV prophylaxis with palivizumab (also known as Synagis), per local standard of care

Key Exclusion Criteria:

1. Previous use of OAV101 or any AAV9 gene therapy
2. Participant with history of aspiration pneumonia or signs of aspiration (eg, coughing or sputtering of food) within 4 weeks prior to Screening
3. Participant dependent on gastrostomy feeding tube for 100% of nutritional intake.
4. Anti-AAV9 antibody titer > 1:50 as determined by ligand binding immunoassay at the time of screening
5. Inability to take corticosteroids
6. Concomitant use of immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, or immunosuppressive therapy within 3 months prior to gene replacement therapy (eg, cyclosporine, tacrolimus, methotrexate, rituximab cyclophosphamide, IV immunoglobulin)
7. Hepatic dysfunction (i.e. AST, ALT, bilirubin, GGT or GLDH, ≥ ULN; CTCAE ≥ 1) at Screening (with the exception of isolated AST elevation: in the absence of other liver laboratory abnormalities, isolated AST elevation is not considered exclusionary)
8. Previously treated with nusinersen (Spinraza®) within 4 months prior to Screening
9. Previously treated with risdiplam (EvrysdiTM) within 15 days prior to Screening (washout period of at least 5 half-lives before Screening)

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Brazil (3):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 participants were enrolled into the study, at five sites from Brazil (three sites) and Argentina (two sites). Six participants were from Argentina and 10 from Brazil.
Pre-assignment Details: On Day -1, participants were admitted to the hospital for pre-treatment baseline procedures including prednisolone treatment per study protocol.
Groups:
- OAV101: A single IV infusion at 1.1e14 vg/kg over approximately 60 minutes
Period: Overall Study
Arm/Group | OAV101
Started | 16
Completed | 14
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | OAV101
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: months]
  Age at dosing | 15.79 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent AEs and SAEs
Description: An AE is any untoward medical occurrence (eg any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Changes from baseline in vital signs, cardiac safety assessments, and clinical laboratory results are reported as Adverse Events if clinically significant and as applicable, per investigator assessment.
Time Frame: Up to Month 18
Population: Full analysis set (FAS) - all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101
Number analyzed (Participants) | 16
Participants
  Any treatment-emergent adverse events | 16
  Any treatment-emergent adverse events related to OAV101 | 11
  Any serious treatment-emergent adverse events | 11
  Serious treatment-emergent adverse events related to OAV101 | 3
  Treatment-emergent adverse events leading to study discontinuation | 0
  Treatment-emergent adverse events leading to death | 2
  Treatment-emergent adverse events of special interest | 12

2. Primary Outcome: Evaluation of Important Identified and Important Potential Risks - Treatment-emergent Adverse Events of Special Interest
Description: An AE is any untoward medical occurrence (eg any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Adverse events of special interest (AESI) are defined by the important identified risk and important potential risk: Hepatotoxicity, Thrombocytopenia, Cardiac adverse events, Sensory abnormalities suggestive of ganglionopathy, and Thrombotic microangiopathy. These were assessed by the investigator.
Time Frame: Up to Month 18
Population: Full analysis set (FAS) - all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101
Number analyzed (Participants) | 16
Participants
  Risk name: Hepatotoxicity | 11
  -Preferred term: Aspartate aminotransferase increased | 5
  -Preferred term: Alanine aminotransferase increased | 5
  -Preferred term: Blood alkaline phosphatase increased | 2
  -Preferred term: Bilirubin conjugated increased | 2
  -Preferred term: Gamma-glutamyltransferase increased | 5
  -Preferred term: Hepatic enzyme increased | 3
  -Preferred term: Hepatic failure | 1
  -Preferred term: Transaminases increased | 2
  Risk name: Thrombocytopenia | 5
  -Preferred term: Platelet count decreased | 4
  -Preferred term: Thrombocytopenia | 1
  Risk name: Thrombotic microangiopathy | 2
  -Preferred term: Thrombotic microangiopathy | 2

3. Secondary Outcome: Number of Participants Who Achieve Development Motor Milestones According to the World Health Organization-Multicentre Growth Reference Study (WHO-MGRS)
Description: The World Health Organization-Multicentre Growth Reference Study (WHO-MGRS) was used to measure developmental motor milestones. This was assessed via the milestone checklist. The 6 developmental milestones are: sitting without support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone and walking alone. A yes response indicates that the patient reached a particular development milestone.
Time Frame: Baseline (Screening), and at Weeks 26, 52 and 78
Population: Full analysis set (FAS) - all treated patients with evaluable assessments at the respective assessment time points.
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101
Number analyzed (Participants) | 16
Participants
  Screening - Sitting without support | 6
  Screening - Hands-and-knees crawling | 2
  Screening - Standing with assistance | 1
  Screening - Walking with assistance | 0
  Screening - Standing alone | 0
  Screening - Walking alone | 0
  Week 26 Sitting without support (n=14): number analyzed (Participants) | 14
  Week 26 Sitting without support (n=14) | 12
  Week 26 Hands-and-knees crawling (n=14): number analyzed (Participants) | 14
  Week 26 Hands-and-knees crawling (n=14) | 2
  Week 26 Standing with assistance (n=14): number analyzed (Participants) | 14
  Week 26 Standing with assistance (n=14) | 2
  Week 26 Walking with assistance (n=14): number analyzed (Participants) | 14
  Week 26 Walking with assistance (n=14) | 2
  Week 26 Standing alone (n=14): number analyzed (Participants) | 14
  Week 26 Standing alone (n=14) | 1
  Week 26 Walking alone (n=14): number analyzed (Participants) | 14
  Week 26 Walking alone (n=14) | 0
  Week 52 Sitting without support (n=13): number analyzed (Participants) | 13
  Week 52 Sitting without support (n=13) | 10
  Week 52 Hands-and-knees crawling (n=13): number analyzed (Participants) | 13
  Week 52 Hands-and-knees crawling (n=13) | 4
  Week 52 Standing with assistance (n=13): number analyzed (Participants) | 13
  Week 52 Standing with assistance (n=13) | 7
  Week 52 Walking with assistance (n=13): number analyzed (Participants) | 13
  Week 52 Walking with assistance (n=13) | 3
  Week 52 Standing alone (n=13): number analyzed (Participants) | 13
  Week 52 Standing alone (n=13) | 6
  Week 52 Walking alone (n=13): number analyzed (Participants) | 13
  Week 52 Walking alone (n=13) | 2
  Week 78 Sitting without support (n=12): number analyzed (Participants) | 12
  Week 78 Sitting without support (n=12) | 10
  Week 78 Hands-and-knees crawling (n=12): number analyzed (Participants) | 12
  Week 78 Hands-and-knees crawling (n=12) | 3
  Week 78 Standing with assistance (n=12): number analyzed (Participants) | 12
  Week 78 Standing with assistance (n=12) | 7
  Week 78 Walking with assistance (n=12): number analyzed (Participants) | 12
  Week 78 Walking with assistance (n=12) | 2
  Week 78 Standing alone (n=12): number analyzed (Participants) | 12
  Week 78 Standing alone (n=12) | 3
  Week 78 Walking alone (n=12): number analyzed (Participants) | 12
  Week 78 Walking alone (n=12) | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the single dose of study treatment plus 18 months post treatment, up to a maximum duration of 18 months.
Groups:
- OAV101A1 1.le 14vg/kg All: A single IV infusion at 1.1e14 vg/kg over approximately 60 minutes
Arm/Group | OAV101A1 1.le 14vg/kg All
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101A1 1.le 14vg/kg All (N=16)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bronchiolitis (Infections and infestations) | 3
COVID-19 (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Renal failure (Renal and urinary disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101A1 1.le 14vg/kg All (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 7
Hypersensitivity (Immune system disorders) | 1
Asymptomatic bacteriuria (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Coxsackie viral infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Bilirubin conjugated increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 5
Hepatic enzyme increased (Investigations) | 3
Platelet count decreased (Investigations) | 4
Transaminases increased (Investigations) | 2
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Irritability (Psychiatric disorders) | 2
Catarrh (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT05073133/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT05073133/SAP_001.pdf